CLINICAL TRIAL: NCT07353567
Title: Long-term Outcomes and Risk Factors of Local Re-Recurrence in Patients With Locally Recurrent Rectal Cancer
Brief Title: Long-term Outcomes and Risk Factors of Local Re-Recurrence in Patients
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cai Zerong, Deputy Director of the Department, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2025ZSLYEC-595
Record Dates: First submitted 2025-12-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Local Re-Recurrence of Malignant Tumor of Rectum; Local Recurrence of Malignant Tumor of Rectum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients without local re-recurrence
- patients with local re-recurrence

SUMMARY:
To analyze the long-term oncological outcome and identify independent risk factors for local re-recurrence in patients undergoing radical salvage surgery for locally recurrent rectal cancer.

DETAILED DESCRIPTION:
Locally recurrent rectal cancer (LRRC) occurs in 5-12% of rectal cancer patients following curative treatment and continues to pose a considerable clinical challenge1-6. At present, radical salvage surgery represents the only potentially curative approach, with 5-year overall survival (OS) rates of 40-55% reported in selected patient cohorts7-11. Despite advances in surgical techniques and systemic treatments, a significant proportion of patients still develops local re-recurrence (LrR) after salvage surgery for LRRC. In a cohort study with a 10 years of follow-up, 42% of LRRC patients undergoing radical surgery developed LrR, with a concomitant distant metastasis rate of 54.8%11, and another multicenter retrospective study reported a 33% rate of LrR12. Nevertheless, data regarding risk factors and the prognosis of LrR remains scarce.

Several clinical factors associated with LrR has been reported, including positive resection margin and the administration of systemic or local treatments13-15. Furthermore, it remains unclear whether clinicopathological characteristics-from the primary tumor through to local recurrence-can predict the risk of re-recurrence after salvage radical resection.

Therefore, this study aimed to investigate the incidence of LrR among LRRC patients who underwent radical salvage surgery at a high-volume tertiary center in China, and to identify independent prognostic factors associated with LrR. The results may contribute to improving postoperative surveillance and facilitating the development of individualized management strategies for LRRC patients.

ELIGIBILITY:
Inclusion Criteria:

* (1). Patients had undergone curative-intent resection for a histologically confirmed primary rectal or rectosigmoid adenocarcinoma. A disease-free interval ≥3 months was required to distinguish subsequent local recurrence from persistent disease;
* (2). LRRC located within the true pelvis or at the pelvic brim, confirmed by radiological imaging (e.g., MRI, CT, PET-CT) and/or pathological verification;
* (3). Patients who underwent radical salvage surgery (R0/R1) for LRRC. No evidence of residual disease or early second recurrence was observed within 3 months after salvage surgery.
* (4). Availability of complete clinicopathological and treatment-related data.

Exclusion Criteria:

* (1). History of synchronous or metachronous other primary malignancies;
* (2). R2 resection for LRRC;
* (3). Presence of uncontrollable synchronous distant metastasis at the time of either primary tumor treatment or LRRC diagnosis;
* (4). Patients lost to follow-up or lacking essential survival data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 284 patients who underwent radical salvage surgery for LRRC were included in the study, from January 1st, 2010 to March 1st, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Local re-recurrence free survival | LrRFS was calculated from the date of salvage radical surgery until the date when any local re-recurrence was detected by imaging or histology, or until censored at the last follow-up or death, assessed up to 180 months.]
post-recurrent overall survival | PROS was calculated from the date of salvage radical surgery until the date of death or until censored at the last follow-up, assessed up to 180 months.

IPD SHARING:
Plan to Share IPD: No
Please contact us by Email